CLINICAL TRIAL: NCT04329780
Title: Retrospective Multicenter Comparison of Laparoscopic and Robotic-Assisted Roux-en-Y Gastric Bypass and Sleeve Gastrectomy
Brief Title: Retrospective Comparison of Lap and Robotic-Assisted RYGB and SG
Status: Completed | Type: Observational
Sponsor: Intuitive Surgical (Industry)
Responsible Party: Sponsor
Other Study IDs: ISI-dVBAR-001
Record Dates: First submitted 2020-03-30; First posted 2020-04-01 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Bariatric Surgery Candidate

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
A retrospective, multicenter, comparative chart review study comparing laparoscopic and robotic-assisted Roux-en-Y Gastric Bypass (RYGB) and Sleeve Gastrectomy (SG)

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older at the time of procedure
* Undergone either laparoscopic or robotic-assisted Roux-en-Y gastric bypass (RYGB) or sleeve gastrectomy (SG)
* Meets qualification for primary bariatric procedure per American Society for Metabolic and Bariatric Surgery guidelines

Exclusion Criteria:

* Subject who underwent bariatric procedure as an emergency procedure
* Subject who underwent bariatric procedure as an revisional bariatric procedure
* Subject who underwent bariatric procedure as an secondary procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who meets all inclusion and exclusion criteria and who have undergone a primary bariatric procedure.
Sampling Method: Non-Probability Sample
Enrollment: 1872 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Perioperative complications | 30 days after surgery
  Peri-operative complications include adverse events during the Intra-operative and post-operative periods.

CONTACTS AND LOCATIONS:
Locations (1):
- Orlando Health, Orlando, Florida, United States